CLINICAL TRIAL: NCT01290081
Title: Prevalence of Latent Tuberculosis and Enhanced Tuberculosis Case Detection Among Injecting Drug Users Receiving Methadone Substitution Treatment
Brief Title: Enhanced Tuberculosis Case Detection Among Substitution Treatment Patients
Acronym: TBIDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Health Development, Estonia (Other Government)
Collaborators: LLC Corrigo (Unknown); Ida-Viru Central Hospital, Department of Tuberculosis (Unknown)
Responsible Party: Kristi Rüütel, National Institute for Health Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TBIDU-1230
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Injecting drug users; Case management
MeSH Terms: conditions — Tuberculosis

ARMS (2):
- Active referral (Active Comparator): Case management intervention group - study personnel scheduled the TB doctor appointment for the participant, reminded to keep it, and transportation to the clinic was organized when needed.
  Interventions: Other: Case management approach in referral to health care services
- Passive referral (No Intervention): Participants were instructed to schedule an appointment with TB services themselves.
  Interventions: Other: Case management approach in referral to health care services

INTERVENTIONS:
Other: Case management approach in referral to health care services — Case management intervention aimed at increasing TB screening and treatment entry among injecting drug users referred from a methadone drug treatment program

SUMMARY:
The purpose of this study was to determine the prevalence of latent tuberculosis infection among injecting drug users and to conduct randomized controlled trial to evaluate a case management intervention aimed at increasing TB screening and treatment entry among injecting drug users referred from a methadone drug treatment program in Estonia.

ELIGIBILITY:
Inclusion Criteria:

* Participation in substitution treatment program,
* Age 18 years or more,
* Able to read and write in Estonian or Russian,
* Able to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- LLC Corrigo, Jõhvi, Ida-Virumaa, Estonia

REFERENCES:
- [Derived] Ruutel K, Loit HM, Sepp T, Kliiman K, McNutt LA, Uuskula A. Enhanced tuberculosis case detection among substitution treatment patients: a randomized controlled trial. BMC Res Notes. 2011 Jun 15;4:192. doi: 10.1186/1756-0500-4-192. PMID 21676222